CLINICAL TRIAL: NCT02837510
Title: Neural Mechanisms Associated With Risk of Smoking Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 824061; 5R01DA041402 (NIH)
Record Dates: First submitted 2016-06-03; First posted 2016-07-19 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Nicotine Addiction
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard smoking cessation counseling (Other): Participants will receive a standard treatment program consisting of smoking cessation counseling.
  Interventions: Behavioral: Standard smoking cessation counseling

INTERVENTIONS:
Behavioral: Standard smoking cessation counseling — Participants will discuss reasons for quitting, the model of smoking as a learned habit, triggers for smoking, and trigger management; receive brief training in how to manage withdrawal symptoms and relapse prevention counseling and receive the NCI Clearing the Air self-help smoking cessation booklet. The target quit date (TQD) session will be scheduled to occur up to 2 weeks following the pre-quit session. Participants will then meet with a smoking cessation counselor for a 15 minute booster counseling session. During the first week following TQD there will be two monitoring visits to closely monitor abstinence. Weekly thereafter for four weeks, participants will attend a brief booster counseling session.

SUMMARY:
This study will examine how abstinence-induced brain changes contribute to smoking cessation outcomes in treatment-seeking smokers.

DETAILED DESCRIPTION:
Smoking is the greatest preventable cause of mortality and a significant economic burden. Even with the best available treatments, most smokers relapse within days or weeks after a quit attempt. Nicotine replacement therapy, the most widely used pharmacotherapy, yields end of treatment quit rates of <25% suggesting that managing nicotine withdrawal is not sufficient. To improve quit rates significantly, a more refined mechanistic understanding is needed. Neuroimaging can identify mechanisms underlying behavior change beyond self-report and behavioral measures. Functional magnetic resonance imaging (fMRI) studies show that brief (e.g., 24 hr.) abstinence from smoking produces working memory deficits associated with reduced neural activity in cognitive control circuits. This study will examine how abstinence-induced brain changes contribute to clinical outcomes in treatment-seeking smokers. Using a validated fMRI abstinence challenge paradigm, 200 treatment-seeking smokers will complete two 1-hour pre-treatment fMRI scans: after smoking satiety and after 24 hours of confirmed abstinence. Approximately 50% of participants will complete the smoking session first, followed by the absence session, and the remainder will complete the opposite order (counterbalanced). The investigators will examine brain responses during the performance of tasks probing working memory. Participants will then set a target quit date, receive smoking cessation counseling, and be monitored for 6 months to assess time to relapse using a validated smoking relapse protocol.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be:

1. Treatment-seeking smokers between the ages of 18 and 65, reporting consumption of at least 5 cigarettes per day for at least the past 6 months;
2. Planning to live in the area for at least the next 3 months;
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form;
4. Able to communicate fluently in English (speaking, writing, and reading).

Exclusion Criteria:

Subjects who present and/or self-report with the following criteria at any point during study participation will not be eligible to participate in the study:

Smoking Behavior:

1. Use of chewing tobacco or snuff or cigars;
2. Current enrollment or plans to enroll in another smoking cessation program or research study in the next 3 months;
3. Current or anticipated (within the next 3 months) use of smoking cessation medications or nicotine replacement therapy (NRT);
4. A baseline carbon monoxide (CO) reading less than or equal to 8ppm.

Alcohol/Drugs:

1. Diagnosis or treatment for alcohol or drug abuse in the past two years as reported during phone screen (e.g., alcohol, opioids, cocaine, or stimulants);
2. Current alcohol consumption that exceeds 25 standard drinks/week;
3. Positive breath alcohol concentration test (BrAC greater than or equal to 0.01) at intake;

   a. Participants testing positive for breath alcohol with a reading equal to or greater than .08 (the legal driving limit) or who are visibly impaired will be instructed not to drive themselves home after the appointment. If a participant needs to use a phone to call for a safe ride home, an office telephone will be made available to the participant.
4. A positive urine drug screen for cocaine, opiates, PCP, benzodiazepines, methadone, MDMA, amphetamine, methamphetamine, tri-cyclic antidepressants and/or barbiturates at any session;

Medication:

Current use or recent discontinuation (within the past 30 days at the time of Intake) of:

1. Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin SR, Chantix, NRT);
2. Anti-psychotic medications;
3. Anti-depressants (tricyclics, SSRI's, selective and nonselective MAOIs, Wellbutrin/Zyban);
4. Anti-anxiety agents;
5. Anti-panic agents;
6. Prescription (e.g., Provigil, Ritalin) or over-the-counter stimulants;
7. Prescription sleep aids (e.g., Ambien, Lunesta) if used more than 2x/week. If participants report use less than twice a week, they will just be asked to refrain from use during imaging portion of the study.
8. Any medication that could compromise participant safety as determined by the Principal Investigator and/or Study Physician;

   Daily use of:
9. Opiate-containing medications for chronic pain.

Medical/Neuropsychiatric:

1. Women who are pregnant, planning a pregnancy, and/or breast feeding. All female subjects of childbearing potential will undergo a urine pregnancy test at Intake and both fMRI scan visits (3 urine pregnancy tests in total).
2. History of epilepsy or a seizure disorder;
3. History of stroke;
4. Self-reported brain or spinal tumor;
5. Self-reported history or current diagnosis of psychosis, bipolar disorder, schizophrenia, current major depression (subjects with a history of major depression but in remission for past 6 months are eligible), or any Axis 1 disorder.

fMRI-Related:

1. Self-reported history of head trauma;
2. Self-reported brain (or CNS) or spinal tumor;
3. Self-reported use of pacemakers, certain metallic implants, or presence of metal in the eye as contraindicated for fMRI;
4. Self-reported history of claustrophobia;
5. Being left-handed;
6. Color blindness;
7. Weight greater than 299lbs;
8. Self-reported history of gunshot wounds;
9. Any impairment preventing participants from using the response pad necessary for the cognitive testing;
10. Circumstances or conditions that may interfere with magnetic resonance imaging (MRI).

General Exclusion:

1. Any medical condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator;
2. Low or borderline intellectual functioning - determined by a score of less than 85 on the Shipley Institute of Living Scale (SILS) (administered at Intake Visit);
3. Enrollment or plans to enroll in another research study;
4. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Loughead, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allenby C, Falcone M, Wileyto EP, Cao W, Bernardo L, Ashare RL, Janes A, Loughead J, Lerman C. Neural cue reactivity during acute abstinence predicts short-term smoking relapse. Addict Biol. 2020 Mar;25(2):e12733. doi: 10.1111/adb.12733. Epub 2019 Feb 25. PMID 30806013
- See also: Click here for more information about this study: Neural mechanisms associated with risk of smoking relapse — http://www.phillyquit.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After study intake participants were randomized to one of two scan order: Abstinent then Smoking, Smoking then Abstinent.
Groups:
- Abstinent Then Smoking: This group received abstinent session first in counterbalanced order.
- Smoking Then Abstinent: This group received smoking session first in counterbalanced order.
Period: 1st Pretreatment fMRI Session
Arm/Group | Abstinent Then Smoking | Smoking Then Abstinent
Started | 61 | 58
Completed | 60 | 57
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Washout (2 Weeks)
Arm/Group | Abstinent Then Smoking | Smoking Then Abstinent
Started | 60 | 57
Completed | 59 | 56
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: 2nd Pretreatment fMRI Session
Arm/Group | Abstinent Then Smoking | Smoking Then Abstinent
Started | 59 | 56
Completed | 58 | 55
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Quit Attempt (6 Months)
Arm/Group | Abstinent Then Smoking | Smoking Then Abstinent
Started | 58 | 55
Completed | 56 | 53
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Standard Smoking Cessation Counseling
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 111
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 72
  White | 35
  More than one race | 5
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 119
Fagerstrom Test For Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Nicotine Dependence is an instrument for assessing the intensity of physical addiction to nicotine. It provides an ordinal measure of nicotine dependence related to cigarette smoking and is composed 6 items measuring the quantity of cigarette consumption, the compulsion to use, and dependence. Yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to produce a total score of 0-10. The higher the total score, the more intense the patient's physical dependence on nicotine.
  units on a scale | 4.72 (1.79)

OUTCOME MEASURES:

1. Primary Outcome: Days to Relapse
Description: The primary outcome will be the number of days to relapse following the target quit date. Relapse will be confirmed using a conventional SRNT guideline criterion of either a positive biochemical verification of smoking or 7 consecutive days of smoking based on self-report (it is very unlikely that a subject would meet the latter criterion without also meeting the former, given the long half-life of cotinine). The days to relapse will be based upon time from target quit date to the first day of the relapse period. Self-reported daily smoking data will be collected using a validated timeline follow-back method. Self-reported abstinence will be biochemically verified on a weekly basis using urine cotinine (<100ng/ml) and a CO reading of ≤5PPM. Drop-outs will be considered relapsers following the last date of abstinence data provided.
Time Frame: 6 months after target quit date
Population: Participants completing both fMRI sessions (smoking, abstinent) and starting the quit period were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abstinent Then Smoking | Smoking Then Abstinent
Number analyzed (Participants) | 58 | 55
days | 3.95 (2.67) | 3.78 (2.69)

2. Secondary Outcome: Brain Activation (BOLD Percent Signal Change)
Description: To measure the effects of acute 24-hour abstinence from smoking on executive function, functional magnetic resonance imaging (fMRI) was utilized to assess the relative importance of dorsolateral prefrontal cortex (left DLPFC, right DLPFC), Medial Frontal/Cingulate Gyrus (MF/CG), Posterior Cingulate Cortex (PCC) and Prefrontal cortex (PFC) blood oxygen dependent (BOLD) signals during working memory task performance. Measurement of BOLD percent signal change range is 0 to 2%. Percent signal change is the difference in fMRI signal between the baseline condition (B) and the task condition (T) and calculated here as: percent signal change = (T-B)/B×100%. Greater percent signal change in the DLPFC, MF/CG, PCC, and PFC is generally associated with better executive function.
Time Frame: 24 hours
Population: Participants completing both fMRI sessions (smoking, abstinent) were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of signal change
Groups:
- Pre-treatment fMRI Abstinent Session: This session was conducted following a 24 hr period of abstinence from smoking.
- Pre-treatment fMRI Smoking Session: This session was conducted following a 24 hr period of smoking as usual.
Arm/Group | Pre-treatment fMRI Abstinent Session | Pre-treatment fMRI Smoking Session
Number analyzed (Participants) | 115 | 115
percentage of signal change
  Left DLPFC | 0.23 (0.349) | 0.26 (0.268)
  RIght DLPFC | 0.22 (.331) | 0.23 (0.240)
  MF/CG | 0.21 (0.307) | 0.24 (0.239)
  PCC | -0.25 (0.306) | -0.34 (0.239)
  PFC | -0.31 (0.491) | -0.37 (0.389)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Pre-treatment fMRI Abstinent Session: Reporting AEs experienced for all participants during the Abstinent session. This session was conducted following a 24 hr period of abstinence from smoking.
- Washout (2 Weeks): A two-week washout period (smoking as usual) separated scan 1 and scan 2.
- Pre-treatment fMRI Smoking Session: Reporting AEs experienced for all participants during the smoking session. This session was conducted following a 24 hr period of smoking as usual.
- Quit Attempt (6 Months): Following the completion of the pretreatment fMRI session, participants set a target quit date, received smoking cessation counseling, and were monitored for six months.
Arm/Group | Pre-treatment fMRI Abstinent Session | Washout (2 Weeks) | Pre-treatment fMRI Smoking Session | Quit Attempt (6 Months)
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/117 | 0/115 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/117 | 0/115 | 4/113
Other Adverse Events (participants affected / at risk) | 0/117 | 1/117 | 1/115 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-treatment fMRI Abstinent Session (N=117) | Washout (2 Weeks) (N=117) | Pre-treatment fMRI Smoking Session (N=115) | Quit Attempt (6 Months) (N=113)
Hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Voluntary hospitalization for psychiatric symptoms.
Hypoglycemic event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hospitalization due to knee replacement
hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant hospitalized for respiratory infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-treatment fMRI Abstinent Session (N=117) | Washout (2 Weeks) (N=117) | Pre-treatment fMRI Smoking Session (N=115) | Quit Attempt (6 Months) (N=113)
vertigo (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accident (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — participant involved in a minor car accident

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT02837510/Prot_SAP_000.pdf